CLINICAL TRIAL: NCT00440115
Title: Disease Management for Smokers in Rural Primary Care
Brief Title: Disease Management for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01CA101963 (NIH); 5R01CA101963 (NIH)
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Bupropion; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- High intensity disease management (Experimental): High intensity disease management, free nicotine replacement therapy or bupropion
  Interventions: Behavioral: High intensity disease management; Drug: Bupropion
- Low intensity disease management (Experimental): Low intensity disease management, free nicotine replacement therapy or bupropion
  Interventions: Behavioral: Low intensity disease management; Drug: Bupropion
- Comparison group (Other): Comparison group, free nicotine replacement therapy or bupropion
  Interventions: Behavioral: Comparison group; Drug: Bupropion

INTERVENTIONS:
Behavioral: High intensity disease management — Health education mailings, 6 motivation interviews/counseling
  Arms: High intensity disease management
Behavioral: Low intensity disease management — Health education mailings, one motivation interview/counseling
  Arms: Low intensity disease management
Behavioral: Comparison group — Health education mailings
  Arms: Comparison group
Drug: Bupropion — Buproprion or Nicotine Replacement Therapy
  Other Names: Nicotine Replacement Therapy

SUMMARY:
The primary aim of this study is to assess the effectiveness of both high and low intensity, disease management programs for smoking. The hypotheses are to compare abstinence from cigarettes, the number of quit attempts, and smokers motivation at 24 months between participants receiving high and low intensity disease management and those receiving usual care.

DETAILED DESCRIPTION:
The primary aim of this study is to assess the effectiveness of both high and low intensity, disease management programs for nicotine dependence. In this study, we will recruit 750 smokers from 20 rural, primary care clinics in Kansas. Subjects will be randomly assigned to one of three study arms, each providing 20 months of treatment: C (comparison group), LDM (low-intensity disease management) or HDM (high-intensity disease management). Participants in group C will receive health educational mailings and an offer for free nicotine replacement therapy (six weeks) or bupropion (seven weeks) every 6 months (months 0, 6, 12, and 18). Participants in LDM will receive the same interventions as C plus a low-intensity disease management program that includes a single telephone counseling session using motivational interviewing (MI) at months 0, 6, 12, and 18 to encourage a cessation attempt and also includes coordination of smoking assessments and pharmacotherapy with the patient's physician. HDM participants will receive C plus a high intensity disease management program that includes up to six telephone-based MI counseling sessions at months 0, 6, 12, and 18 to encourage a smoking cessation attempt and to prevent relapse after a quit attempt, as well as coordination of smoking assessments, quit attempts, and pharmacotherapy with the patient's physician.

The primary outcome of the study is 7-day point prevalence abstinence from cigarettes at 2 years after enrollment. Secondary outcomes include: 1) number of quit attempts and 2) progress in stage of change. If successful, this intervention will provide a generalizable model for addressing nicotine dependence that could improve long-term management of smoking in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Reported smoking at least 10 cigarettes per day for at least 25 of the last 30 days
* Speak English
* Their regular physician is a participating physician
* Working home telephone or cellular phone

Exclusion Criteria:

* Women who are pregnant or planning to become pregnant in the next two years
* Plan on moving within two years
* Display signs of dementia or other mental disorders
* Live with a smoker already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. Ellerbeck, MD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Result] Cox LS, Wick JA, Nazir N, Cupertino AP, Mussulman LM, Ahluwalia JS, Ellerbeck EF. Predictors of early versus late smoking abstinence within a 24-month disease management program. Nicotine Tob Res. 2011 Mar;13(3):215-20. doi: 10.1093/ntr/ntq227. Epub 2011 Jan 13. PMID 21233256
- [Result] Cupertino AP, Wick JA, Richter KP, Mussulman L, Nazir N, Ellerbeck EF. The impact of repeated cycles of pharmacotherapy on smoking cessation: a longitudinal cohort study. Arch Intern Med. 2009 Nov 9;169(20):1928-30. doi: 10.1001/archinternmed.2009.355. PMID 19901150
- [Result] Ellerbeck EF, Mahnken JD, Cupertino AP, Cox LS, Greiner KA, Mussulman LM, Nazir N, Shireman TI, Resnicow K, Ahluwalia JS. Effect of varying levels of disease management on smoking cessation: a randomized trial. Ann Intern Med. 2009 Apr 7;150(7):437-46. doi: 10.7326/0003-4819-150-7-200904070-00003. PMID 19349629
- [Result] Cox LS, Cupertino AP, Mussulman LM, Nazir N, Greiner KA, Mahnken JD, Ahluwalia JS, Ellerbeck EF. Design and baseline characteristics from the KAN-QUIT disease management intervention for rural smokers in primary care. Prev Med. 2008 Aug;47(2):200-5. doi: 10.1016/j.ypmed.2008.04.013. Epub 2008 May 3. PMID 18544464
- [Result] Berg CJ, Sanderson Cox L, Mahnken JD, Greiner KA, Ellerbeck EF. Correlates of self-efficacy among rural smokers. J Health Psychol. 2008 Apr;13(3):416-21. doi: 10.1177/1359105307088144. PMID 18420774
- [Result] Hutcheson TD, Greiner KA, Ellerbeck EF, Jeffries SK, Mussulman LM, Casey GN. Understanding smoking cessation in rural communities. J Rural Health. 2008 Spring;24(2):116-24. doi: 10.1111/j.1748-0361.2008.00147.x. PMID 18397444
- [Result] Cupertino PA, Richter KP, Cox LS, Nazir N, Greiner AK, Ahluwalia JS, Ellerbeck EF. Smoking cessation pharmacotherapy preferences in rural primary care. Nicotine Tob Res. 2008 Feb;10(2):301-7. doi: 10.1080/14622200701825817. PMID 18236294
- [Result] Cupertino AP, Mahnken JD, Richter K, Cox LS, Casey G, Resnicow K, Ellerbeck EF. Long-term engagement in smoking cessation counseling among rural smokers. J Health Care Poor Underserved. 2007 Nov;18(4 Suppl):39-51. doi: 10.1353/hpu.2007.0117. PMID 18065851
- [Result] Berg CJ, Cox LS, Nazir N, Mussulman LM, Ahluwalia JS, Ellerbeck EF. Correlates of home smoking restrictions among rural smokers. Nicotine Tob Res. 2006 Jun;8(3):353-60. doi: 10.1080/14622200600670132. PMID 16801293
- [Derived] Yeh HW, Ellerbeck EF, Mahnken JD. Simultaneous evaluation of abstinence and relapse using a Markov chain model in smokers enrolled in a two-year randomized trial. BMC Med Res Methodol. 2012 Jul 7;12:95. doi: 10.1186/1471-2288-12-95. PMID 22770436

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Smokers screened for eligibility (n=1827)
  Ineligible (n=714)
  Invited to participate (n=1113)
  Declined to participate (n=305) Unable to contact (n=58)
  Randomly assigned (n=750)
Groups:
- High-intensity Disease Management: Health education mailings, free nicotine replacement therapy or bupropion, 6 motivational interviewing/counseling sessions
- Moderate-intensity Disease Management: Health education mailings, free nicotine replacement therapy or bupropion, 2 motivational interviewing/counseling sessions
- Pharmacotherapy Management (Comparison Group): Health education mailings, free nicotine replacement therapy or bupropion
Period: Overall Study
Arm/Group | High-intensity Disease Management | Moderate-intensity Disease Management | Pharmacotherapy Management (Comparison Group)
Started | 251 | 249 | 250
Completed | 244 | 238 | 244
Not Completed | 7 | 11 | 6
Not completed — Death | 7 | 9 | 5
Not completed — Incarceration | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-intensity Disease Management | Moderate-intensity Disease Management | Pharmacotherapy Management (Comparison Group) | Total
Number analyzed (Participants) | 251 | 249 | 250 | 750
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.5) | 48.2 (12.4) | 47.1 (13.4) | 47.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 144 | 144 | 439
  Male | 100 | 105 | 106 | 311
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 4 | 12
  Not Hispanic or Latino | 249 | 243 | 246 | 738
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 2 | 7
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 2 | 8
  White | 221 | 225 | 225 | 671
  More than one race | 19 | 18 | 19 | 56
  Unknown or Not Reported | 1 | 3 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 251 | 249 | 250 | 750
Stage of change [Count of Participants; unit: Participants]
  Precontemplation | 23 | 20 | 22 | 65
  Contemplation | 146 | 153 | 158 | 457
  Preparation | 82 | 76 | 70 | 228

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Abstinence From Cigarettes
Description: Self-reported 7-day point prevalence abstinence from cigarettes
Time Frame: 24 months
Population: We used generalized linear models for the primary endpoint (self-reported abstinence at 24 months). Missing values were imputed as smokers, deaths and incarcerations were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High-intensity Disease Management | Moderate-intensity Disease Management | Pharmacotherapy Management (Comparison Group)
Number analyzed (Participants) | 244 | 238 | 244
Participants | 68 | 56 | 56
Statistical Analysis 1: Comparison: High-intensity Disease Management vs Moderate-intensity Disease Management vs Pharmacotherapy Management (Comparison Group); Test type: Superiority — Power calculations demonstrated that 250 participants per group would have 95% power to compare combined high-intensity disease management and moderate-intensity disease management with pharmacotherapy management, on the basis of 10% (pharmacotherapy management), 15% (moderate-intensity disease management), and 25% (high-intensity disease management) self-reported quit rates; p = 0.54, Mixed Models Analysis; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.78 to 1.61] — (High-intensity disease management and moderate-intensity disease management) vs pharmacotherapy management
Statistical Analysis 2: Comparison: High-intensity Disease Management vs Moderate-intensity Disease Management; Test type: Superiority — Power calculations indicated that 250 participants per group would have 80% power to compare high-intensity disease management and moderate-intensity disease management with pharmacotherapy management, on the basis of 10% (pharmacotherapy management), 15% (moderate-intensity disease management), and 25% (high-intensity disease management) self-reported quit rates; p = 0.18, Mixed Models Analysis; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.88 to 2.02] — High-intensity disease management vs moderate-intensity disease management

2. Secondary Outcome: Number of Quit Attempts
Description: Number of quit attempts at 6, 12, 18, and 24 months. A quit attempt is defined as use of quit-smoking pharmacotherapy (nicotine patch or bupropion) during each treatment period.
Time Frame: 6, 12, 18, 24 months
Measure: Number; unit: quit attempts
Arm/Group | High-intensity Disease Management | Moderate-intensity Disease Management | Pharmacotherapy Management (Comparison Group)
Number analyzed (Participants) | 251 | 249 | 250
quit attempts
  Month 6 : Quit Attempted | 171 | 160 | 142
  Month 6 : Deceased/Incarcerated | 2 | 4 | 3
  Month 6 : No Quit Attempt | 78 | 85 | 105
  Month 12 : Quit Attempted | 95 | 93 | 114
  Month 12 : Deceased/Incarcerated | 3 | 5 | 3
  Month 12 : No Quit Attempt | 153 | 151 | 133
  Month 18 : Quit Attempted | 61 | 49 | 65
  Month 18 : Deceased/Incarcerated | 6 | 9 | 3
  Month 18 : No Quit Attempt | 184 | 191 | 182
  Month 24 : Quit Attempted | 59 | 65 | 55
  Month 24 : Deceased/Incarcerated | 7 | 11 | 6
  Month 24 : No Quit Attempt | 185 | 173 | 189

3. Secondary Outcome: Progress in Stage of Change
Description: Progress in Stages of Change at 6, 12, 18, and 24 months
Time Frame: 6, 12, 18, 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | High-intensity Disease Management | Moderate-intensity Disease Management | Pharmacotherapy Management (Comparison Group)
Number analyzed (Participants) | 251 | 249 | 250
Participants
  Month 6: Pre-contemplation | 24 | 25 | 15
  Month 6: Contemplation | 65 | 74 | 89
  Month 6: Preparation | 87 | 84 | 98
  Month 6: Quit (Action/Maintenance) | 43 | 37 | 28
  Month 6: Unknown | 30 | 25 | 17
  Month 6: Deceased/Incarcerated | 2 | 4 | 3
  Month 12: Pre-contemplation | 25 | 34 | 24
  Month 12: Contemplation | 70 | 71 | 83
  Month 12: Preparation | 50 | 57 | 79
  Month 12: Quit (Action/Maintenance) | 59 | 50 | 38
  Month 12: Unknown | 44 | 32 | 23
  Month 12: Deceased/Incarcerated | 3 | 5 | 3
  Month 18: Pre-contemplation | 23 | 31 | 17
  Month 18: Contemplation | 55 | 67 | 81
  Month 18: Preparation | 44 | 44 | 74
  Month 18: Quit (Action/Maintenance) | 63 | 49 | 44
  Month 18: Unknown | 60 | 49 | 31
  Month 18: Deceased/Incarcerated | 6 | 9 | 3
  Month 24: Pre-contemplation | 30 | 32 | 33
  Month 24: Contemplation | 59 | 61 | 70
  Month 24: Preparation | 31 | 37 | 46
  Month 24: Quit (Action/Maintenance) | 81 | 65 | 66
  Month 24: Unknown | 43 | 43 | 29
  Month 24: Deceased/Incarcerated | 7 | 11 | 6

ADVERSE EVENTS:
Arm/Group | High-intensity Disease Management | Moderate-intensity Disease Management | Pharmacotherapy Management (Comparison Group)
All-Cause Mortality (participants affected / at risk) | 7/251 | 11/249 | 6/250
Serious Adverse Events (participants affected / at risk) | 15/251 | 2/249 | 2/250
Other Adverse Events (participants affected / at risk) | 63/251 | 46/249 | 19/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-intensity Disease Management (N=251) | Moderate-intensity Disease Management (N=249) | Pharmacotherapy Management (Comparison Group) (N=250)
Dystonia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial Surgery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibriliation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Broken Neck (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bronchitis/COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Collapsed lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — As a result of a rodeo injury
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Depression and Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Kidney Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Removal of Lung Mass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Smoke Inhalation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — As a result of occupational hazard
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Surgery (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-intensity Disease Management (N=251) | Moderate-intensity Disease Management (N=249) | Pharmacotherapy Management (Comparison Group) (N=250)
Chest Pain (Product Issues) | 0 (0) | 3 (3) | 1 (1)
Cold Sores (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Constipation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Depression (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Dizziness/Light Headedness (Product Issues) | 1 (1) | 3 (3) | 1 (1)
Elevated heart rate or blood pressure (Product Issues) | 3 (3) | 6 (6) | 1 (1)
Flu (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Headache (Product Issues) | 0 (0) | 4 (4) | 0 (0)
Blood Clot (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Bowel Falure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Broken Bone (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — As a result of a fall
Crohn's Disease Complication (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes Complication (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1) | 2 (2)
Shingles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Strep Throat (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scheduled Surgery/Medical Procedure (Surgical and medical procedures) | 9 (9) | 3 (3) | 1 (1)
Irritability/Nervousness (Product Issues) | 1 (1) | 2 (2) | 3 (3)
Nausea (Product Issues) | 5 (5) | 7 (7) | 1 (1)
Nose Bleeds (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Shakiness (Product Issues) | 2 (2) | 3 (3) | 0 (0)
Skin Irritation (Product Issues) | 15 (15) | 8 (8) | 7 (7)
Sleep Disturbance (Product Issues) | 4 (4) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No